CLINICAL TRIAL: NCT05048329
Title: The Cascade Feasibility Pilot (Ileostomy): Improving Care Processes for New Ileostomy Patients Using Continuous Remote Patient Monitoring and a Cascading Alert System
Brief Title: The Cascade Feasibility Pilot (Ileostomy)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Endeavor Health (Other)
Responsible Party: Principal Investigator, Nirav Shah, Medical Director of Quality Innovation and Clinical Practice Analytics, Program Director of Outcomes Research for Quality and Transformation, Endeavor Health
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: EH20-288 Cascade Ileostomy
Record Dates: First submitted 2021-09-08; First posted 2021-09-17 (Actual); Results first posted 2024-05-21 (Actual); Last update posted 2024-05-21 (Actual); Status verified 2024-05

CONDITIONS: Ileostomy; Complications; Ileostomy - Stoma
Keywords: Ileostomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ileostomy Cohort (Experimental): The study will include ten eligible patients into the cohort to conduct the study.
  Interventions: Other: Non-invasive continuous remote monitoring with structured escalation pathway; Other: Affective Analysis of Participant Response to Continuous Remote Patient Monitoring

INTERVENTIONS:
Other: Non-invasive continuous remote monitoring with structured escalation pathway — Continuous patient monitoring through non-invasive biosensors coupled with machine learning algorithms, with a structured escalation and communication pathway for home health providers and colorectal clinical team
Other: Affective Analysis of Participant Response to Continuous Remote Patient Monitoring — Surveys and interviews with enrolled participants

SUMMARY:
Existing interventions including improving communication and self-care to improve readmission of patients undergoing high risk colorectal surgery involving new ileostomy formation has shown limited results. Our proposal is to deploy a wearable solution that predicts physiological perturbation with continuous remote patient monitoring and advanced machine learning algorithms which will be connected to structured, cascading, escalation pathways and care coordination involving home health nurses, colorectal and ostomy nurses, and colorectal surgeons, and has the potential to transform surgical management in the post-discharge period, where patients are the most vulnerable for readmission. This feasibility study will contribute to the understanding of post-discharge continuous remote monitoring of ileostomy patients, promote patient self-care, and has the potential of improving patient outcomes.

DETAILED DESCRIPTION:
Colorectal surgery is a high-risk surgery that results in significant morbidity, and health care utilization in the form of readmission. Ileostomy creation is a significant risk factor in colorectal surgery rehospitalization. Effective continuous remote patient monitoring (CRPM) can reduce readmissions, but it has only been realized in select heart failure populations via invasive monitoring. The investigators will focus on colorectal CRPM in the elective, new ileostomy population through a structured cascading and escalating alert system. In this feasibility study, the investigators will use a wearable biosensor and collect ambulatory physiological data that are analyzed by machine learning algorithms, to generate personalized alerts of physiological perturbation in colorectal surgery patients in the post-discharge period. Alerts from this algorithm may be cascaded with other patient status data to inform management by the home health team via a structured protocol built into the electronic health record (EHR). The escalation pathway will engage home health nurses, colorectal care team nurses, ostomy nurses, and colorectal surgeons. The investigators will conduct surveys and semi-structured interviews with patients, and semi-structured interviews with providers, which will be used to evaluate the perceptions, acceptance, and experience of this CRPM solution.

ELIGIBILITY:
Inclusion Criteria:

* Patient is inpatient admission at NorthShore University HealthSystem hospital
* Patient underwent a new ileostomy formation at index hospitalization
* Patient is at least 18 years of age
* Patient is fluent in English
* Patient agrees to protocol-required procedures
* Patient discharges with NorthShore Home Health Service

Exclusion Criteria:

* Patient has cognitive or physical limitations that, in the investigator's opinion, limit the patient's ability to maintain patch device and phone
* Patient has allergy to hydrocolloid adhesives
* Patient has present skin damage preventing them from wearing a study device
* Pregnancy
* Patient discharge location is a Skilled Nursing Facility or other subacute facilities

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2021-08-09 (Actual); Primary Completion 2022-05-31 (Actual); Study Completion 2022-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nirav S Shah, Principal Investigator — Endeavor Health
Locations (3):
- United States (3):
  - NorthShore University HealthSystem Evanston Hospital, Evanston, Illinois
  - NorthShore University HealthSystem Glenbrook Hospital, Glenview, Illinois
  - NorthShore University HealthSystem HighlandPark Hospital, Highland Park, Illinois

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment was conducted at three NorthShore Hospitals from August 2021 and September 2022
Pre-assignment Details: A total of 11 participants were enrolled in the study. One patient withdrew and one was a screen fail, resulting in a total of 9 participants who completed the study.
Groups:
- Ileostomy Cohort: The study will include 10 eligible patients into the study cohort to conduct the study.
Period: Overall Study
Arm/Group | Ileostomy Cohort
Started | 11
Completed | 9
Not Completed | 2
Not completed — Withdrawal by Subject | 1
Not completed — Screenfail | 1

BASELINE CHARACTERISTICS:
Population: The number of participants completed the study
Arm/Group | Ileostomy Cohort
Number analyzed (Participants) | 9
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 6
  >=65 years | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 9
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 7
  More than one race | 0
  Unknown or Not Reported | 2

OUTCOME MEASURES:

1. Primary Outcome: Attrition Rate
Description: Drop out from study
Time Frame: 30 days from patient discharge date
Measure: Count of Participants; unit: Participants
Arm/Group | Ileostomy Cohort
Number analyzed (Participants) | 11
Participants | 2

2. Primary Outcome: Enrollment Rate
Description: Enrollment rate for entire patient cohort
Time Frame: Through study completion, an average of 30 days for each patient
Measure: Count of Participants; unit: Participants
Arm/Group | Ileostomy Cohort
Number analyzed (Participants) | 23
Participants | 11

3. Secondary Outcome: 30 Days Readmission
Description: 30-day readmission to hospital
Time Frame: 30 days from patient discharge date
Measure: Count of Participants; unit: Participants
Arm/Group | Ileostomy Cohort
Number analyzed (Participants) | 9
Participants | 1

4. Secondary Outcome: Number of Participants With Stool Regimen Escalation
Description: Frequency of stool regimen escalation by providers
Time Frame: 30 days from patient discharge date
Measure: Count of Participants; unit: Participants
Arm/Group | Ileostomy Cohort
Number analyzed (Participants) | 9
Participants | 2

ADVERSE EVENTS:
Time Frame: We collected adverse event data over the 30-day participation period for each participant
Arm/Group | Ileostomy Cohort
All-Cause Mortality (participants affected / at risk) | 0/11
Serious Adverse Events (participants affected / at risk) | 0/11
Other Adverse Events (participants affected / at risk) | 0/11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol (2023-03-08): https://cdn.clinicaltrials.gov/large-docs/29/NCT05048329/Prot_000.pdf